CLINICAL TRIAL: NCT02316769
Title: Randomized Controlled Trial Comparing the McGrath MAC Video Laryngoscope With the King Vision Video Laryngoscope in Adult Patients.
Brief Title: Comparison Study of the McGrath MAC Video Laryngoscope With the King Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Bret Alvis, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120884
Record Dates: First submitted 2014-09-05; First posted 2014-12-15 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2016-07

CONDITIONS: Video Laryngoscopic Device Usage in Novice Users

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- King Vision Video Laryngoscope (Active Comparator): Patient intubated with the King Vision Video Laryngoscope
  Interventions: Procedure: King Vision video laryngoscope
- McGrath MAC Video Laryngoscope (Active Comparator): Patient intubated with the McGrath MAC Video Laryngoscope
  Interventions: Procedure: McGrath MAC video laryngoscope

INTERVENTIONS:
Procedure: King Vision video laryngoscope — Patient intubated with the King Vision Video Laryngoscope
  Arms: King Vision Video Laryngoscope
Procedure: McGrath MAC video laryngoscope — Intubation with the McGrath MAC video laryngoscope
  Arms: McGrath MAC Video Laryngoscope

SUMMARY:
In this study, the investigators compare the effectiveness of two relatively new video laryngoscopes, McGrath MAC (Covidien, Dublin Ireland) and the King Vision (King Systems, Noblesville, IN), by practitioners experienced in airway management but with limited exposure to these two devices. Our hypothesis was that, the McGrath MAC device would require fewer intubation attempts and shorter intubation times than the King Vision when performed by novice users.

ELIGIBILITY:
Inclusion Criteria:

* All interested airway providers (Residents, Attendings, Certified Nurse Anesthetist and
* Student Registered Nurse Anesthetist) will be eligible to be included. -

Exclusion Criteria:

* All patients with difficult airways as determined by history or physical exam (limited oral opening, limited cervical extension, receding chin, Mallampati class III or IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Alvis, Principal Investigator — Vanderbilt University

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the King Vision arm one patient was removed from the surgery secondary to a planned procedure change and another was removed from the study because they declined to participate after already signing consent for this study. This explains the 31 patient enrollment in the King Vision arm.
Groups:
- King Vision Video Laryngoscope: Patient intubated with the King Vision Video Laryngoscope
  Intubation with the King Vision video laryngoscope
Period: Overall Study
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope
Started | 33 | 33
Completed | 31 | 33
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (15) | 52 (21) | 52 (17)
Sex/Gender, Customized [Number; unit: participants]
  Male | 18 | 15 | 33
  Female | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Intubation Success on First Attempt as Measured by End Tidal Carbon Dioxide
Time Frame: participants were followed up to the point the video device is removed from the airway, classified as under 90 seconds.
Measure: Number; unit: participants
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope
Number analyzed (Participants) | 31 | 33
participants | 24 | 33

2. Secondary Outcome: Time to Intubation
Description: Number of patients intubated in less than 90 seconds
Time Frame: Intubation time was initiated at the time of entry of the study device beyond the teeth/gum line and the intubation time was stopped when the study device was removed beyond the same point.
Measure: Number; unit: participants
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope
Number analyzed (Participants) | 31 | 33
participants | 10 | 25

ADVERSE EVENTS:
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No